CLINICAL TRIAL: NCT06756698
Title: The Intervention Effect and Potential Neural Mechanisms of Music Therapy in Children and Adolescents with NSSI
Brief Title: The Intervention Effect and Potential Neural Mechanisms of Music Therapy in Children and Adolescents with Mood Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-07
Record Dates: First submitted 2024-12-10; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-07

CONDITIONS: Mood Disorders in Children and Adolescents
Keywords: NSSI; music therapy; children and adolescent; mood disorders; hyperscanning
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional treatment (Active Comparator): The conventional treatment group receives DBT group therapy 5 times a week, each time for 1 hour, and also received individual personalized therapy twice a week.
  Interventions: Other: conventional treatment
- conventional treatment plus music intervention (Experimental): The music therapy group receives individual music therapy twice a week, 30 minutes each time, for a total of 3 weeks on top of conventional treatment.
  Interventions: Other: conventional treatment plus music intervention

INTERVENTIONS:
Other: conventional treatment plus music intervention — Each music therapy session will include 5 stages. In stage 1, an emotional assessment is conducted to observe the patient's current emotional experience and feelings (provide a VAD score), which lasts about 1 minute. In stage 2, relaxation exercises (breathing relaxation, progressive muscle relaxation, and imaginary relaxation) are conducted under the guidance of the therapist to the music corresponding to the relaxation target VAD, which lasts about 8 minutes. In stage 3, the patient independently selects the music and discusses it with the therapist, which lasts about 10 minutes. In stage 4, the patient listens to resource and positive-oriented music and discusses specific topics with the therapist, which lasts about 10 minutes. Finally, in stage 5, the therapist again conducts an emotional assessment of the patient and observes the patient's current emotional experience and feelings, which lasts about 1 minute.
  Arms: conventional treatment plus music intervention
Other: conventional treatment — The conventional treatment group received DBT group therapy 5 times a week, each session lasting 1 hour, and also received individual personalized therapy twice a week.
  Arms: conventional treatment

SUMMARY:
This study plans to combine questionnaires, scales, electrophysiological and neuroimaging methods to comprehensively evaluate the effectiveness of music therapy for children and adolescents with emotional disorders and NSSI, and explore the potential neural mechanisms of its effectiveness.

DETAILED DESCRIPTION:
The subjects will be randomly divided into the conventional treatment group (TAU) and the music therapy group (MT). The conventional treatment group will receive DBT group therapy 5 times a week, 1 hour each time, and individual personalized therapy twice a week; the music therapy group will receive individual music therapy twice a week, 30 minutes each time, for a total of 3 weeks on top of conventional treatment.

During each intervention, near-infrared brain functional imaging, electrodermal and electrocardiographic equipment will be used to synchronously collect multimodal data from therapists and patients. The heart rate variability, electrodermal conductance response of therapists and patients, and the relative concentrations of oxygenated hemoglobin (oxy-Hb), deoxyhemoglobin (deoxy-Hb) and total hemoglobin in the brain tissue of the subjects and therapists were monitored during the treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed;
* Born and raised in China, with Chinese as the only native language;
* Voluntary participation, with the consent of the family members of patients under 18 years old, and signed the informed consent form;
* Meet the diagnostic criteria of DSM-5 anxiety disorder or depressive disorder;
* There have been two or more self-harm behaviors in the past six months.

Exclusion Criteria:

* Meet the diagnostic criteria of DSM-5 psychotic disorder, manic episode, autism spectrum disorder, mental retardation, tic disorder, substance abuse and other mental illnesses;
* Severe organic brain disease;
* Hearing loss or loss of music-related pleasure;
* Those who have clear suicidal ideation, attempt and behavior in the past month.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
psychological scale measurement：Screen for Child Anxiety Related Emotional Disorders (SCARED) | before and after three weeks of music intervention
  Before and after the entire music intervention course, Screen for Child Anxiety Related Emotional Disorders (SCARED) scale is administered to the subjects as baseline and final data. The minimum value is 0. The maximum value is 82. Higher scores means a worse result(the more anxious the person is). A total score of ≥ 25 may indicate the presence of an Anxiety Disorder. Scores higher than 30 are more specific.
psychological scale measurement：Beck Depression Inventory-II (BDI-II) | before and after three weeks of music intervention
  Before and after the entire music intervention course, Beck Depression Inventory-II (BDI-II) scale is administered to the subjects as baseline and final data. This scale is used to assess the severity of depressive symptoms in the past two weeks, and contains 21 items, each item is scored on a level of 0~3, and the total score of the scale is the sum of the scores of 21 items. According to the cut-off score provided by the original scale such as Beck, the total score of 0~13 is no depression, 14~19 is mild depression, 20~28 is moderate depression, and 29~63 is severe depression. The minimum value is 0. The maximum value is 63. Higher scores means a worse result.
psychological scale measurement：Beck Scale for Suicide Ideation (BSS) | before and after three weeks of music intervention
  Before and after the entire music intervention courseBeck Scale for Suicide Ideation (BSS) scale is administered to the subjects as baseline and final data. There are 3 options for the scale answers, and the corresponding scores from left to right are 1, 2, and 3, with the higher the score, the stronger the desire to die. All visitors complete the first 5 questions first, and if the answer to the 4th and 5th items is "no", then they are considered to have no suicidal ideation and complete this questionnaire; If any one of the 4th or 5th items is "weak" or "moderate to strong", then it is considered suicidal ideation and you need to continue to complete the next 14 items. The higher the score, the greater the intensity of suicidal ideation. Higher scores means a worse result.

SECONDARY OUTCOMES:
psychological scale measurement：Children's Depression Inventory (CDI) | before and after three weeks of music intervention
  Before and after the entire music intervention course, Children's Depression Inventory (CDI) scale is administered to the subjects as baseline and final data. The minimum value is 0. The maximum value is 54. Higher scores means a worse result.
psychological scale measurement：Fear of Negative Evaluation Scale (FNE) | before and after three weeks of music intervention
  Before and after the entire music intervention course, Fear of Negative Evaluation Scale (FNE) scale is administered to the subjects as baseline and final data. The scale is scored from 12 to 60. The opposite of a high FNE is the absence of concern about the evaluation of others, as opposed to the expectation or need for a positive evaluation.
psychological scale measurement：Emotion Regulation Questionnaire (ERQ) | before and after three weeks of music intervention
  Before and after the entire music intervention course, Emotion Regulation Questionnaire (ERQ) scale is administered to the subjects as baseline and final data. The Emotion Regulation Questionnaire is designed to assess individual differences in the habitual use of two emotion regulation strategies: cognitive reappraisal and expressive suppression. There are 2 parts of the score, the higher of each score means the more the person use this strategy.
psychological scale measurement：Alexian Brothers Urge to Self-Injure Scale (ABUSI) | before and after three weeks of music intervention
  Before and after the entire music intervention course, Alexian Brothers Urge to Self-Injure Scale (ABUSI) scale is administered to the subjects as baseline and final data. The Alexian Brothers Urge to Self-Injure Scale (ABUSI) assesses the motivation of an individual to engage in self-injury. The minimum value is 0. The maximum value is 35. Higher scores means a worse result.
psychological scale measurement：Difficulties in Emotion Regulation Scale (DERS) | before and after three weeks of music intervention
  Before and after the entire music intervention course, Difficulties in Emotion Regulation Scale (DERS) scale is administered to the subjects as baseline and final data. The DERS is a brief, 36-item self-report questionnaire designed to assess multiple aspects of emotional dysregulation. The measure yields a total scorev(SUM) as well as scores on six sub-scales: 1. Non-acceptance of emotional responses (NONACCEPT); 2. Difficulties engaging in goal directed behaviour (GOALS ); 3. Impulse control difficulties (IMPULSE); 4. Lack of emotional awareness (AWARE); 5. Limited access to emotion regulation strategies (STRATEGIES); 6. Lack of emotional clarity (CLARITY). Higher scores suggest greater problems with emotion regulation.
psychological scale measurement：Center for Epidemiologic Studies Depression Scale (CES-D) | before and after three weeks of music intervention
  Before and after the entire music intervention course, Center for Epidemiologic Studies Depression Scale (CES-D) scale is administered to the subjects as baseline and final data. The minimum value is 0. The maximum value is 20. Higher scores means a worse result. The total score of ≤15 points is no depressive symptoms, 16~19 points are possible depressive symptoms, and ≥ 20 points are definitely depressive symptoms.
DBT-Ways of Coping Checklist (DBT-WCCL) | before and after three weeks of music intervention
  The Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL) was designed to assess participants' use of DBT skills (e.g., acceptance, cognitive reappraisal, problem-solving) and maladaptive coping responses (e.g., avoidance, denial, self-blame). This is a 59-item self-report scale where participants rate their use of the scale with a four-point scale, resulting in two subscales: a DBT Skills Subscale (DSS) and a Dysfunctional Coping Subscale (DCS).
  The scoring is the average of relevant items for each subscale. The score for the skills use scale is the average of these items: 1, 2, 4, 6, 9, 10, 11, 13, 16, 18, 19, 21, 22, 23, 26, 27, 29, 31, 33, 34, 35,36, 38, 39, 40, 42, 43, 44, 47,49, 50, 51, 53, 54, 56, 57, 58,59 The dysfunctional coping scale 1 (general dysfunctional coping factor) has these items: 3,5, 8, 12, 14,17, 20, 25, 32, 37, 41, 45, 46,52, 55 and the dysfunctional coping scale 2 (blaming others factor) has these items: 7,15, 24, 28, 30,48

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to the restrictions outlined in the participants' informed consent, data are available upon request.